CLINICAL TRIAL: NCT03727867
Title: A Randomized Ⅲ Phase Trial of Efficacy of Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Combined With Early Stereotactic Body Radiation Therapy to the Primary Tumor in Advanced Non-small Cell Lung Cancer Patients Harboring Epidermal Growth Factor Receptor Mutation
Brief Title: Efficacy of Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Combined With Early Stereotactic Body Radiation Therapy to the Primary Tumor in Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Haihua Yang (Other)
Responsible Party: Sponsor-Investigator, Haihua Yang, the head of radiotherapy department in Taizhou Hospital, Taizhou Hospital
Organization: Taizhou Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Target-SBRT
Record Dates: First submitted 2018-10-27; First posted 2018-11-01 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Advanced Non-small Cell Lung Cancer
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug group (Placebo Comparator): Participants were under prescription of Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR TKI) at the beginning and continued until disease progressed.
  Interventions: Drug: Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor
- Drug plus SBRT group (Experimental): After the first month of EGFR TKI orally, participants were given Stereotactic Body Radiation Therapy (SBRT) in dose of 50 Gy/5 F or 60 Gy/8 F for peripheral and central primary tumor, respectively, combined with oral EGFR TKI continually until the primary end point.
  Interventions: Drug: Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor; Device: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor — Oral EGFR TKI begins on day 1 and continues until disease progresses.
  Other Names: EGFR TKI
Device: Stereotactic Body Radiation Therapy — Participants were given Stereotactic Body Radiation Therapy in a dose of 60 Gy/8 fraction for the central tumor or 50 Gy/5 fraction for the peripheral lung cancer, respectively.
  Other Names: SBRT; stereotactic ablative radiotherapy (SABR)
  Arms: Drug plus SBRT group

SUMMARY:
Non-small cell lung cancer (NSCLC) is a prevalent disease with high mortality and morbidity, particularly of adenocarcinoma in Asians. Fortunately, with the development of epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor (TKI), treatment of lung cancer usher in a new era, resulting in a hit of precise therapy and molecule sequencing. However, it is inevitable for patients to gain acquired resistance of EGFR TKI. Several studies have been demonstrated that there were approximately 30% heterogeneous cells in primary tumors. And emerging studies illuminated that main pattern of treatment failure was the recurrence of primary site. Moreover, it was proved that despite of the drug-resistance cells in progressive site, continual prescription of EGFR TKI in oligometastasis lung cancer could make a difference for patients in progression free survival (PFS) and overall survival (OS), owing to the residual responsive cells in another sites. Therefore, to explore an unique method to control heterogeneous cells in primary site so as to delay or prevent acquired resistance when taking EGFR TKI orally may be of great benefit and therapy.

It is known to all that stereotactic body radiation therapy (SBRT), with the advantage of hypofractionation and rapid release, succeed in several cancers, such as early lung cancer, prostatic, liver cancer and so on, for local control. Numerous reports explained SBRT played an irreplaceable role in progressive NSCLC patients after oral targeted medicine, regardless of EGFR or anaplastic lymphoma kinase (ALK) mutation. And the radiosensitivity of EGFR TKI in vitro and vivo may account for these inspiring results. What's more, it has reported that SBRT could induce inflammatory cell death, activate dendritic cell as well as accelerate antigen presentation in the draining lymph node, leading to antigen-specific adaptive immune response. Nevertheless, although the potential effects of SBRT on advanced NSCLC are obviously, few studies explore the preventive benefits of early SBRT combined with oral EGFR TKI on advanced lung cancer by eliminating the heterogeneous cells in primary site. In addition, the investigators' previous phase II study of SBRT combined with oral EGFR TKI had revealed its safety and potentially improvement of PFS for 6 months.

In this trial, the investigators put sight into assessing the efficacy of early application of SBRT to primary site in the advanced NSCLC patients and provide a hypothesis that early SBRT could strengthen the anti-tumor effect of EGFR TKI through eradicating the heterogenity of initial tumor cells.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must sign a study specific informed consent form prior to clinical trial;
2. World Healthy Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2 and kamofsky performance status (KPS) >60 at enrollment;
3. Patients must have tumors that were proven histopathologically or cytologically as advanced non-small cell lung cancer and that harbored sensitizing EGFR mutation (e.g. exon 19 deletion or exon 21 L858R);
4. Estimated life expectancy >8 weeks;
5. Patients should have adequate bone marrow function defined as absolute peripheral granulocyte count (AGC) of >/= 1500 cells/mm3, platelet count of >/= 100000 cells/mm3; adequate hepatic function with bilirubin </= 1.5 mg/dl, creatinine clearance >/= 50 ml/min and international normalized ration (INR) 0.8-1.2; adequate lung function: forced expiratory ration in 1 second >80%;
6. The number of oligometastasis plus primary lesion should be less that 5, and the maximum diameter of the primary lesion in lung should be under 5 cm, without tracheal and thoracic vessels invasion.

Exclusion Criteria:

1. Patients must be withdrawn with prior radiotherapy, chemotherapy, immunotherapy and surgery of chest;
2. Uncontrolled intercurrent illness including but not limited to, ongoing or active infection, failure in bone marrow, liver, kidney, heart and lung, or psychiatric illness/social situations that would limit compliance with study requirements;
3. Patients who suffered from symptomatic intracranial metastasis or other malignant tumors, such as cervical cancer,skin cancer and so on;
4. Patients who participated other clinical drug trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Duration of time from the start of EGFR TKI therapy to the time of disease progression, assessed up to 3 years.
  Evaluate the effect of EGFR TKI with or without SBRT on progression free survival.

SECONDARY OUTCOMES:
Local control rate (LCR) | Up to 3 years.
  To describe the rate of local control and out-of-field disease progression, irrespectively.
Overall survival | Duration of time from the start of EGFR TKI therapy to 3 years or until time of death, whichever occurs first.
  To evaluate overall survival in EGFR TKI therapy with SBRT in comparison to EGFR TKI therapy alone.
Adverse events | Up to 3 years.
  The acute and chronic profile associated with the study regimen using CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Hailing Xu, MM, Principal Investigator — Taizhou Hospital, Wenzhou Medical University
Locations (1):
- Taizhou Hospital, Wenzhou Medical University, Taizhou, Zhejiang, China